CLINICAL TRIAL: NCT01853657
Title: Efficacy of First and Second Line ART in HIV Patients Treated at the Komfo Anokye Teaching Hospital, Kumasi
Brief Title: Kumasi Cohort Study
Acronym: KCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bernhard Nocht Institute for Tropical Medicine (Other Government)
Collaborators: Kwame Nkrumah University of Science and Technology (Other); Kumasi Centre for Collaborative Research (KCCR) (Other); Komfo Anokye Teaching Hospital (Other); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Kirsten A. Eberhardt, Dr., MD, Bernhard Nocht Institute for Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KCS
Record Dates: First submitted 2013-05-08; First posted 2013-05-15 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Virological monitoring (Active Comparator): In addition to routine clinical and immunological monitoring with CD4 counts
  Interventions: Other: Virological monitoring
- Routine monitoring (No Intervention): Immunological and clinical monitoring

INTERVENTIONS:
Other: Virological monitoring
  Arms: Virological monitoring

SUMMARY:
The main objective is to access efficacy of first and second line antiretroviral therapy (ART) and its determinants in patients treated at the Komfo Anokye Teaching Hospital in Kumasi (KATH), Ghana, and to compare the clinical, virological and immunological efficacy of second line ART in patients who were switched after virological failure compared to patients who were switched after clinical or immunological failure.

Other specific study objectives are:

1. To establish an HIV Cohort Study at the study site.
2. To assess the rate of virological failure among patients on first line therapy
3. To compare the clinical, immunological and virological efficacy of second line antiretroviral therapy amongst patients randomised to virological monitoring whilst on first line compared with those monitored routinely using clinical and immunological monitoring.
4. To assess the incidence and outcome of tuberculosis (TB) and other opportunistic infections in patients treated at the Komfo Anokye Teaching Hospital HIV services
5. To obtain parameters for quality of care, e. g. performance of TB screening procedures
6. To develop strategies to minimise treatment failures, on the basis of the results of the study
7. To generate a large prospective second-line ART cohort, to serve as basis for further research projects
8. To implement point-of-care viral load analysis at the Komfo Anokye Teaching Hospital
9. Capacity building: epidemiology, medical documentation and data base management. Enrollment of one PhD and one Master student

DETAILED DESCRIPTION:
Study design:

Open randomized study

Recruitment:

All patients being on stable ART for at least one year will be asked to participate in the study after thorough information about the objectives/procedures of the study and associated inconveniences/risks. After informed consent has been given, patients will be asked to complete a short questionnaire on their history of antiretroviral therapy, including information on drug adherence, reliability of drug supply, side effects and complications of highly active antiretroviral therapy (HAART). Data on the socioeconomic status, perceived difficulties related to antiretroviral therapy and subjective quality of care and support offered by the HIV treatment program will be documented.

Randomization:

Patients will be randomized to arm I (n=1500), with viral load testing (VL) in addition to clinical and immunological monitoring according to the algorithm listed below, or to group II (all other eligible patients, at least n=1500), with clinical and immunological monitoring (CI) only. Randomization will be conducted according to a computer list.

Blood sampling:

In addition to the blood drawn for the routine workup of HIV services (CD4 cell count, biochemistry), an additional 10ml blood sample (5ml EDTA, 5ml serum) will be obtained from all patients enrolled in the study for analysis of viral load and major confounders for ART outcome, as e. g. viral hepatitis. Additionally, a blood sample (5ml EDTA plasma) will be taken from patients in the arm II (CI) before switching to second line ART upon clinical or immunological failure for viral load analysis.

Viral load analysis:

To assure timely clinical availability of viral load testing, point of care testing is required and shall be established at KATH. A Cobas® Amplicore Analyzer (Roche Diagnostics) has been installed at KATH but is not routinely used, although functional, due to lacking resources. Viral load testing shall be conducted after adequate training of staff and servicing of the machine has been assured.

Definition of therapy failure:

Therapy failure will be defined according to WHO and national guidelines for antiretroviral therapy:

1. Clinical failure is the occurrence of a new opportunistic infection or malignancy signifying clinical disease progression, the recurrence of prior opportunistic infection or onset/recurrence of WHO stage 3 or 4 conditions.
2. Immunologic failure is the return of CD4 counts to pre-therapy baseline, or below and/or more than 50% fall from on-therapy CD4 peak-level (and/or more than 50% fall in CD4), or persistent low CD4 of less than 100 cells/µl after one year of therapy without other concomitant infection to explain the low CD4.
3. Virological failure is defined as plasma HIV-1 RNA level above 5,000 copies/mL in a person who has been on a regimen for more than 6 months without other concomitant infection to explain the rise or non-suppression of the viral load and in whom drug adherence is determined to be sufficient.

In patients with viral load > 5000 copies per mL and evidence of insufficient drug adherence, adherence counseling is conducted and viral load is controlled after 3 months. If viral load is again > 5000 copies per mL, and adherence is determined to be sufficient, patients shall be switched to second line ART. In patients with a viral load between 50 and 5,000 copies per mL, adherence counseling is conducted and viral load is repeated between 3 to 6 months. Patients with a viral load >500 copies per mL upon control shall be switched to second-line ART.

ART Switch:

Patients who meet the definition of virological, immunological or clinical failure as specified above, will be informed about the indication to switch to second-line ART according to national guidelines, about the benefit and possible side effects second-line ART. Patients however have the choice to refuse being switched to second-line treatment. Currently, recommended and available second-line regimes are:

1. Tenofovir plus lamivudine for patients failing a first line backbone of zidovudine plus lamivudine or
2. Zidovudine plus lamivudine for patients failing a backbone of Tenofovir plus lamivudine together with Lopinavir/ritonavir.

Other available backbone available but seldom used include Abacavir and didanosine.

Adherence monitoring and counseling:

Adherence is monitored by self reporting, pill counts and pharmacy records, as indicated in the national guidelines for antiretroviral therapy. All patients with virological, immunological or clinical therapy failure will receive adherence counseling before switching to second-line ART. Patients with detectable viral load will equally receive adherence counseling, before controlling viral load after 3 months.

Follow-up:

Patients are re-evaluated according to national guidelines. Patients without detectable viral load or evidence for treatment failure will be seen every 6 months or more frequently if clinically indicated. Patients who are switched to second-line ART will be closely followed up to assess tolerance. Usually, this is within 14 days after initiation of treatment, then monthly for the first 3 month, and then in intervals of 2-6 months.

End points:

Primary end point:

Combined endpoint is clinical failure 12 and 24 months after switch to second line treatment, defined as:

1. First/new AIDS defining event
2. Death

Secondary end points:

1. Absolute number of CD4 cells at the diagnosis of therapy failure
2. Mean increase in CD4 cell count after 12/24months
3. Frequency and time of therapy changes, Lost-to-follow up
4. ART-related Adverse Events (AE)
5. Adherence

Interventions:

Apart from viral load analysis in a subgroup of randomly assigned patients, no interventions are carried out within this study. Viral load results will be made available to clinicians treating patients to help in their management.

Sample size calculation:

No substantiated data have been reported regarding the expected difference in the combined primary endpoint, the occurrence of clinical failure (death or new AIDS defining event) after switch to second line ART between the groups. Based on existing data, we assume an incidence of the primary endpoint of about 4% in the first year after switch to second line ART [1]. To detect a difference of 1.5% after a follow-up period of one year with a power of 0.8, a sample size of 626 patients (313 per group) is needed. By screening 1500 patients with viral load testing, with an assumed rate of virological failure of 30%, a total of 450 patients will be offered second line ART [2]. Thus, assuming that 20-30% of those will either not give informed consent, drop out or will be not evaluable, it appears adequate to randomize and 1500 patients for viral load analysis to achieve the calculated sample size.

Statistical analysis:

An interim analysis will be done for primary and secondary end points 12 and 24 months after recruitment is completed. Because the number of patients with clinical failure becoming evident during the recruitment period will be lower than the number of patients with treatment failure detected by viral load analysis, patients having being already started on second-line ART upon clinical failure will be evaluated retrospectively.

Statistical analysis will be performed using the SPSS statistics 19 software package.

ELIGIBILITY:
Inclusion Criteria:

* able and willing to give informed written consent
* age > 18 years
* on first line ART since > 12 months

Exclusion Criteria:

* not willing or able to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2012-06; Primary Completion 2021-06-28 (Actual); Study Completion 2021-07-28 (Estimated)

PRIMARY OUTCOMES:
Clinical failure | 12 and 24 months
  Combined endpoint is clinical failure 12 and 24 months after switch to second line treatment, defined as:
  1. First/new AIDS defining event
  2. Death

SECONDARY OUTCOMES:
CD4 response | 12 and 24 months
  Absolute number of CD4 cells at the diagnosis of therapy failure and mean increase in CD4 cell count after 12 or 24 months

OTHER OUTCOMES:
Frequency and time of therapy changes | 12 and 24 months
Loss-to-follow up | 12 and 24 months
ART-related Adverse Events (AE) | 12 and 24 months
Adherence | 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Fred S Sarfo, FWACP, PHD, Principal Investigator — Kwame Nkrumah University of Science and Technology; Kirsten A Eberhardt, Dr., MD, Principal Investigator — Bernhard Nocht Institute for Tropical Medicine
Locations (1):
- Komfo Anokye Teaching Hospital, Kumasi, Ghana

REFERENCES:
- [Background] Keiser O, Tweya H, Braitstein P, Dabis F, MacPhail P, Boulle A, Nash D, Wood R, Luthi R, Brinkhof MW, Schechter M, Egger M; ART-LINC of IeDEA Study Group. Mortality after failure of antiretroviral therapy in sub-Saharan Africa. Trop Med Int Health. 2010 Feb;15(2):251-8. doi: 10.1111/j.1365-3156.2009.02445.x. Epub 2009 Dec 9. PMID 20003034
- [Background] Seyler C, Adje-Toure C, Messou E, Dakoury-Dogbo N, Rouet F, Gabillard D, Nolan M, Toure S, Anglaret X. Impact of genotypic drug resistance mutations on clinical and immunological outcomes in HIV-infected adults on HAART in West Africa. AIDS. 2007 May 31;21(9):1157-64. doi: 10.1097/QAD.0b013e3281c615da. PMID 17502726